CLINICAL TRIAL: NCT04665856
Title: A Phase III, Randomized, Double-Blind, Placebo-Controlled Study of Atezolizumab Plus Carboplatin and Etoposide With or Without Tiragolumab in Patients With Untreated Extensive-Stage Small Cell Lung Cancer
Brief Title: Study of Atezolizumab Plus Carboplatin and Etoposide With or Without Tiragolumab in Participants With Untreated Extensive-Stage Small Cell Lung Cancer
Acronym: SKYSCRAPER-02C
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: YO42373
Record Dates: First submitted 2020-12-07; First posted 2020-12-14 (Actual); Results first posted 2025-10-29 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Small Cell Lung Carcinoma
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Tiragolumab; atezolizumab; Carboplatin; Etoposide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Tiragolumab + Atezolizumab + Carboplatin and Etoposide (Experimental): Induction treatment with tiragolumab plus atezolizumab and CE will be administered on a 21-day cycle for 4 cycles. Following the induction phase, participants will continue maintenance therapy with tiragolumab plus atezolizumab for 21-day cycles.
  Interventions: Drug: Tiragolumab; Drug: Atezolizumab; Drug: Carboplatin; Drug: Etoposide
- Placebo + Atezolizumab + Carboplatin and Etoposide (Placebo Comparator): Induction treatment with placebo plus atezolizumab and CE will be administered on a 21-day cycle for 4 cycles. Following the induction phase, participants will continue maintenance therapy with placebo plus atezolizumab for 21-day cycles
  Interventions: Drug: Atezolizumab; Drug: Carboplatin; Drug: Etoposide; Drug: Tiragolumab Matching Placebo

INTERVENTIONS:
Drug: Tiragolumab — Tiragolumab at a fixed dose of 600 milligrams (mg), administered by intravenous (IV) infusion, every 3 weeks (Q3W) on Day 1 of each 21-day cycle.
  Other Names: MTIG7192A
  Arms: Tiragolumab + Atezolizumab + Carboplatin and Etoposide
Drug: Atezolizumab — Atezolizumab at a fixed dose of 1200 mg, administered by IV infusion, Q3W on Day 1 of each 21-day cycle.
  Other Names: Tecentriq
Drug: Carboplatin — Carboplatin administered IV to achieve an initial target area under the concentration time curve (AUC) of 5 mg/mL/min, Q3W on Day 1 of each 21-day cycle for 4 cycles.
Drug: Etoposide — Etoposide 100 mg/m^2, administered by IV infusion, Q3W on Day 1, 2 and 3 of each 21-day cycle for 4 cycles.
Drug: Tiragolumab Matching Placebo — Matching placebo, administered by IV infusion, Q3W on Day 1 of each 21-day cycle.
  Arms: Placebo + Atezolizumab + Carboplatin and Etoposide

SUMMARY:
The purpose of this multicenter study in China is to evaluate the safety and efficacy of tiragolumab plus atezolizumab and carboplatin and etoposide (CE) compared with placebo plus atezolizumab and CE in participants with untreated extensive-stage small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
* Histologically or cytologically confirmed Extensive-Stage Small Cell Lung Cancer (ES-SCLC) per the modified Veterans Administration Lung Study Group (VALG) staging system
* No prior systemic treatment for ES-SCLC
* For participants who have received prior chemoradiotherapy for limited-stage SCLC must have had treatment with curative intent and a treatment-free interval of at least 6 months between the last dose/cycle of chemotherapy, thoracic radiotherapy, or chemoradiotherapy and the diagnosis of ES-SCLC
* Measurable diseases as defined by RECIST v1.1
* Submission of a pre-treatment tumor tissue sample
* Adequate hematologic and end-organ function
* Participants not receiving therapeutic anticoagulation with International Normalized Ratio (INR) and Activated Clotting Time (aPTT) </= 1.5 x ULN
* Participants receiving therapeutic anticoagulation: stable anticoagulant regimen
* Negative Human Immunodeficiency Virus (HIV) test at screening
* Negative hepatitis B surface antigen (HBsAg) test at screening
* Positive hepatitis B surface antibody (HBsAb) test at screening, or negative HBsAb at screening accompanied by either of the following: negative total hepatitis B core antibody (HBcAb) and/or positive total HBcAb test followed by a negative hepatitis B virus (HBV) DNA test
* Negative hepatitis C virus (HCV) antibody test at screening, or positive HCV antibody test followed by a negative HCV RNA test
* Negative Epstein-Barr virus (EBV) viral capsid antigen (VCA) IgM test or negative EBV polymerase chain reaction (PCR) test at screening
* For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraception, and agreement to refrain from donating eggs
* For men: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive methods, and agreement to refrain from donating sperm.

Exclusion Criteria:

* Symptomatic or actively progressing central nervous system (CNS) metastases
* Spinal cord compression
* Leptomeningeal disease
* Uncontrolled pleural effusion, pericardial effusion, or ascites
* Uncontrolled or symptomatic hypercalcemia
* Known clinically significant liver disease, including active viral, alcoholic, or other hepatitis, cirrhosis, and inherited liver disease, or current alcohol abuse
* Malignancies other than SCLC within 5 years prior to randomization
* Active or history of autoimmune disease or immune deficiencies
* History of idiopathic pulmonary fibrosis, organizing pneumonia, drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis on screening chest Computer Tomography (CT) scan
* Known active tuberculosis, Current treatment with anti-viral therapy for HBV or HCV
* Severe chronic or active infection
* Treatment with therapeutic oral or IV antibiotics
* Significant cardiovascular disease
* Major surgical procedure other than for diagnosis
* Prior allogeneic bone marrow transplantation or solid organ transplant
* Any other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition
* Administration of a live, attenuated vaccine
* Prior treatment with CD137 agonists, T-cell co-stimulating, or immune checkpoint blockade therapies
* Treatment with systemic immunostimulatory agents
* Treatment with systemic immunosuppressive medications
* History of severe allergic anaphylactic reactions to chimeric or humanized antibodies or fusion proteins
* Known hypersensitivity to Chinese Hamster Ovary (CHO) cell products or to any component of the tiragolumab or atezolizumab formulations
* History of allergic reactions to carboplatin or etoposide
* Pregnancy or breastfeeding, or intention of becoming pregnant during study treatment or within 5 months after the final dose of atezolizumab or within 90 days after the final dose of tiragolumab or for 6 months after the final dose of carboplatin or etoposide.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2020-12-21 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2026-06-30 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (16):
- China (16):
  - Beijing Cancer Hospital, Beijing
  - Beijing Chest Hospital, Beijing
  - the First Affiliated Hospital of Bengbu Medical College, Bengbu
  - the First Hospital of Jilin University, Changchun
  - Fujian Provincial Cancer Hospital, Fuzhou
  - Cancer Center of Guangzhou Medical University, Guangzhou
  - Sir Run Run Shaw Hospital, School of Medicine, Zhejiang University, Hangzhou
  - Zhejiang Cancer Hospital, Hangzhou
  - Harbin Medical University Cancer Hospital, Harbin
  - The 1st Affiliated Hospital of Nanchang Unversity, Nanchang
  - Shanghai Chest Hospital, Shanghai
  - Zhongshan Hospital Fudan University, Shanghai
  - Fudan University Shanghai Cancer Center, Shanghai
  - Cancer Hospital of Shantou University Medical College, Shantou
  - Wuhan Union Hospital Tongji Medical College, Huazhong University of Science and Technology, Wuhan
  - Henan Cancer Hospital, Zhengzhou

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 17 investigative sites in China. This study is still ongoing.
Pre-assignment Details: A total of 123 participants were randomized in the study in a 1:1 ratio to receive tiragolumab plus atezolizumab and carboplatin + etoposide (CE) or placebo plus atezolizumab and CE. One participant from the tiragolumab arm did not receive tiragolumab and hence was included in the placebo arm group for safety analysis.
Groups:
- Placebo + Atezolizumab + Carboplatin + Etoposide: Participants received atezolizumab, 1200 milligrams (mg), followed by tiragolumab matching placebo, and carboplatin, at a dose targeting initial target area under the concentration-time curve (AUC) of 5 milligrams per mililiter per minute (mg/mL/min) as an intravenous (IV) infusion, once every 3 weeks (Q3W), on Day 1 of each 21-day cycle along with etoposide, 100 milligrams per square meter (mg/m^2), as an IV infusion on Days 1, 2 and 3 of each 21-day cycle for 4 cycles as induction treatment. (1 Cycle = 21 days). Participants then received maintenance treatment with atezolizumab, 1200 mg, followed by tiragolumab matching placebo given as an IV infusion, Q3W, from Day 1 of Cycle 5 until disease progression, loss of clinical benefit, unacceptable toxicity, or symptomatic deterioration attributed to disease progression.
- Tiragolumab + Atezolizumab + Carboplatin + Etoposide: Participants received atezolizumab, 1200 mg, tiragolumab, 600 mg, and carboplatin, at a dose targeting initial target AUC of 5 mg/mL/min as an IV infusion, Q3W, on Day 1 along with etoposide, 100 mg/m^2, as an IV infusion on Days 1, 2 and 3 of each 21-day cycle for 4 cycles as induction treatment. (1 Cycle = 21 days). Participants then received maintenance treatment with atezolizumab, 1200 mg, followed by tiragolumab, 600 mg, given as an IV infusion, Q3W, from Day 1 of Cycle 5 until disease progression, loss of clinical benefit, unacceptable toxicity, or symptomatic deterioration attributed to disease progression.
Period: Overall Study
Arm/Group | Placebo + Atezolizumab + Carboplatin + Etoposide | Tiragolumab + Atezolizumab + Carboplatin + Etoposide
Started | 62 | 61
Safety Evaluable Set (Safety Evaluable Set included all randomized participants who received at least one dose of study treatment.) | 63 (1 participant enrolled in the tiragolumab arm did not receive any dose of tiragolumab and was moved to the placebo arm for safety analysis.) | 60 (1 participant enrolled in the tiragolumab arm did not receive any dose of tiragolumab and was moved to the placebo arm for safety analysis.)
Completed | 0 | 0
Not Completed | 62 | 61
Not completed — Site Terminated by Sponsor | 1 | 0
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Lost to Follow-up | 3 | 2
Not completed — Death | 39 | 44
Not completed — Ongoing in study | 17 | 15

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) included all randomized participants whether or not the participants received the assigned study treatment.
Groups:
- Placebo + Atezolizumab + Carboplatin + Etoposide: Participants received atezolizumab, 1200 mg, followed by tiragolumab matching placebo, and carboplatin, at a dose targeting initial target AUC of 5 mg/mL/min as an IV infusion, Q3W, on Day 1 of each 21-day cycle along with etoposide, 100 mg/m^2, as an IV infusion on Days 1, 2 and 3 of each 21-day cycle for 4 cycles as induction treatment. (1 Cycle = 21 days). Participants then received maintenance treatment with atezolizumab, 1200 mg, followed by tiragolumab matching placebo given as an IV infusion, Q3W, from Day 1 of Cycle 5 until disease progression, loss of clinical benefit, unacceptable toxicity, or symptomatic deterioration attributed to disease progression.
- Total: Total of all reporting groups
Arm/Group | Placebo + Atezolizumab + Carboplatin + Etoposide | Tiragolumab + Atezolizumab + Carboplatin + Etoposide | Total
Number analyzed (Participants) | 62 | 61 | 123
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.9 (8.0) | 62.0 (7.8) | 61.4 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 16
  Male | 54 | 53 | 107
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 62 | 61 | 123
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 62 | 61 | 123
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Investigator-Assessed Progression-Free Survival (PFS) in the Primary Analysis Set (PAS)
Description: PFS was defined as time from randomization to the first occurrence of disease progression (PD), as assessed by the investigator using Response Evaluation Criteria in Solid Tumors, Version 1.1 (RECIST v1.1), or death from any cause, whichever occurs first. PD was defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum of diameters at prior timepoints (including baseline), in addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 millimeters (mm).
Time Frame: Up to 32.3 months
Population: Primary Analysis Set (PAS) included all randomized participants without presence or history of brain metastases at baseline.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo + Atezolizumab + Carboplatin + Etoposide | Tiragolumab + Atezolizumab + Carboplatin + Etoposide
Number analyzed (Participants) | 56 | 54
months | 5.39 [4.30 to 6.77] | 5.59 [4.53 to 7.89]
Statistical Analysis 1: Comparison: Placebo + Atezolizumab + Carboplatin + Etoposide vs Tiragolumab + Atezolizumab + Carboplatin + Etoposide; Test type: Superiority; p = 0.0348, Log Rank — This study is a bridging study without formal testing, the p value here is descriptive; Hazard Ratio (HR) = 0.65, 95% CI 2-sided [0.43 to 0.97]

2. Primary Outcome: Overall Survival (OS) in the PAS
Description: OS was defined as the time from the date of randomization to the date of death from any cause.
Time Frame: Up to 32.3 months
Population: PAS included all randomized participants without presence or history of brain metastases at baseline.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo + Atezolizumab + Carboplatin + Etoposide | Tiragolumab + Atezolizumab + Carboplatin + Etoposide
Number analyzed (Participants) | 56 | 54
months | 13.54 [10.35 to 22.44] | 18.69 [14.26 to 20.86]
Statistical Analysis 1: Comparison: Placebo + Atezolizumab + Carboplatin + Etoposide vs Tiragolumab + Atezolizumab + Carboplatin + Etoposide; Test type: Superiority; p = 0.6105, Log Rank — This study is a bridging study without formal testing, the p value here is descriptive; Hazard Ratio (HR) = 0.89, 95% CI 2-sided [0.56 to 1.40]

3. Secondary Outcome: PFS in the FAS
Description: PFS was defined as time from randomization to the first occurrence of PD, as assessed by the investigator using RECIST v1.1, or death from any cause, whichever occurs first. PD was defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum of diameters at prior timepoints (including baseline), in addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.
Time Frame: Up to 32.3 months
Population: FAS included all randomized participants whether or not the participants received the assigned study treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo + Atezolizumab + Carboplatin + Etoposide | Tiragolumab + Atezolizumab + Carboplatin + Etoposide
Number analyzed (Participants) | 62 | 61
months | 5.39 [4.30 to 6.08] | 5.59 [4.47 to 7.89]
Statistical Analysis 1: Comparison: Placebo + Atezolizumab + Carboplatin + Etoposide vs Tiragolumab + Atezolizumab + Carboplatin + Etoposide; Test type: Superiority; p = 0.1044, Log Rank; Hazard Ratio (HR) = 0.73, 95% CI 2-sided [0.49 to 1.07]

4. Secondary Outcome: OS in the FAS
Description: OS was defined as the time from the date of randomization to the date of death from any cause.
Time Frame: Up to 32.3 months
Population: FAS included all randomized participants whether or not the participants received the assigned study treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo + Atezolizumab + Carboplatin + Etoposide | Tiragolumab + Atezolizumab + Carboplatin + Etoposide
Number analyzed (Participants) | 62 | 61
months | 14.88 [10.68 to 22.44] | 17.31 [12.48 to 20.37]
Statistical Analysis 1: Comparison: Placebo + Atezolizumab + Carboplatin + Etoposide vs Tiragolumab + Atezolizumab + Carboplatin + Etoposide; Test type: Superiority; p = 0.9363, Log Rank; Hazard Ratio (HR) = 0.98, 95% CI 2-sided [0.64 to 1.52]

5. Secondary Outcome: Investigator-Assessed Confirmed Objective Response Rate (ORR) in the PAS
Description: ORR was defined as the percentage of participants with either a confirmed complete response (CR) or partial response (PR) on two consecutive occasions ≥4 weeks apart as assessed by investigator according to RECIST v.1.1. CR was defined as disappearance of all target lesions and any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 millimeters (mm). PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters in the absence of CR. Percentages have been rounded off.
Time Frame: Up to 32.3 months
Population: PAS included all randomized participants without presence or history of brain metastases at baseline.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo + Atezolizumab + Carboplatin + Etoposide | Tiragolumab + Atezolizumab + Carboplatin + Etoposide
Number analyzed (Participants) | 56 | 54
percentage of participants | 58.9 [45.01 to 71.63] | 81.5 [68.13 to 90.30]
Statistical Analysis 1: Comparison: Placebo + Atezolizumab + Carboplatin + Etoposide vs Tiragolumab + Atezolizumab + Carboplatin + Etoposide; Test type: Superiority; p = 0.0136, Chi-square with Schouten Correction; Difference in Overall Response Rates = 22.55, 95% CI 2-sided [4.12 to 39.03]

6. Secondary Outcome: Investigator-Assessed Confirmed ORR in the FAS
Description: ORR was defined as the percentage of participants with either a confirmed CR or PR on two consecutive occasions ≥4 weeks apart as assessed by investigator according to RECIST v.1.1. CR was defined as disappearance of all target lesions and any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters in the absence of CR. Percentages have been rounded off.
Time Frame: Up to 32.3 months
Population: FAS included all randomized participants whether or not the participants received the assigned study treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo + Atezolizumab + Carboplatin + Etoposide | Tiragolumab + Atezolizumab + Carboplatin + Etoposide
Number analyzed (Participants) | 62 | 61
percentage of participants | 59.7 [46.46 to 71.70] | 77.0 [64.20 to 86.46]
Statistical Analysis 1: Comparison: Placebo + Atezolizumab + Carboplatin + Etoposide vs Tiragolumab + Atezolizumab + Carboplatin + Etoposide; Test type: Superiority; p = 0.0493, Chi-square with Schouten Correction; Difference in Overall Response Rates = 17.37, 95% CI 2-sided [-0.22 to 33.60]

7. Secondary Outcome: Investigator-Assessed Duration of Response (DOR) in the PAS
Description: DOR was defined as the time interval from the date of the first occurrence of a confirmed objective response until the first date of PD as determined by the investigator using RECIST v1.1 or death from any cause, whichever occurs first. DOR was evaluated for participants who had an objective response of CR or PR. CR was defined as the disappearance of all target lesions and any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters. PD was defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum of diameters at prior timepoints (including baseline), in addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.
Time Frame: Up to 32.3 months
Population: PAS included all randomized participants without presence or history of brain metastases at baseline. Overall number analyzed is the number of participants with objective response i.e., responders.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo + Atezolizumab + Carboplatin + Etoposide | Tiragolumab + Atezolizumab + Carboplatin + Etoposide
Number analyzed (Participants) | 33 | 44
months | 5.45 [3.91 to 5.95] | 5.52 [4.11 to 8.54]

8. Secondary Outcome: Investigator-Assessed DOR in the FAS
Description: as for outcome 7
Time Frame: Up to 32.3 months
Population: FAS included all randomized participants whether or not the participants received the assigned study treatment. Overall number analyzed is the number of participants with objective response i.e., responders.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo + Atezolizumab + Carboplatin + Etoposide | Tiragolumab + Atezolizumab + Carboplatin + Etoposide
Number analyzed (Participants) | 37 | 47
months | 5.45 [3.91 to 6.14] | 5.55 [4.17 to 7.92]

9. Secondary Outcome: Investigator-Assessed PFS Rates at 6 Months and 12 Months in the PAS
Description: PFS = time from randomization to the first occurrence of PD, per investigator per RECIST v1.1/ death from any cause, whichever occurs first. PFS rate at 6 and 12 = the percentage of participants who have not experienced PD per investigator per RECIST v1.1/ death from any cause at 6 and 12 months. PD =at least a 20% increase in the sum of diameters of target lesions, taking as reference the SOD at prior timepoints (including baseline), in addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. Kaplan-Meier (K-M) method was used to estimate PFS rate. Percentages have been rounded off. Abbreviation used in Statistical Analysis section - Event Free Rate - EFR. The event free rate (for example the inv-PFS free rate of 10.24% at 12-months) used the K-M approach to estimate, which accounts for the censoring, the specific nature of time-to-event data. Naive calculation based on patient proportion will introduce bias.
Time Frame: Month 6, Month 12
Population: PAS included all randomized participants without presence or history of brain metastases at baseline. Overall number analyzed is the number of participants with data available for analysis. Number analyzed is the number of participants with data available at the specified timepoint.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo + Atezolizumab + Carboplatin + Etoposide | Tiragolumab + Atezolizumab + Carboplatin + Etoposide
Number analyzed (Participants) | 21 | 25
percentage of participants
  Month 6 | 39.11 [26.09 to 52.14] | 47.20 [33.76 to 60.64]
  Month 12: number analyzed (Participants) | 5 | 14
  Month 12 | 10.24 [1.91 to 18.57] | 27.69 [15.51 to 39.87]
Statistical Analysis 1: Comparison: Placebo + Atezolizumab + Carboplatin + Etoposide vs Tiragolumab + Atezolizumab + Carboplatin + Etoposide; 6 Months; Test type: Superiority; p = 0.3968, Z-test; Difference in EFR at Month 6 = 8.09, 95% CI 2-sided [-10.62 to 26.81]
Statistical Analysis 2: Comparison: Placebo + Atezolizumab + Carboplatin + Etoposide vs Tiragolumab + Atezolizumab + Carboplatin + Etoposide; 12 Months; Test type: Superiority; p = 0.0205, Z-test; Difference in EFR at Month 12 = 17.45, 95% CI 2-sided [2.69 to 32.21]

10. Secondary Outcome: Investigator-Assessed PFS Rates at 6 Months and 12 Months in the FAS
Description: PFS was defined as time from randomization to the first occurrence of PD, as assessed by the investigator using RECIST v1.1, or death from any cause, whichever occurs first. PFS rate at 6 months and 12 months defined as the percentage of participants who have not experienced PD as determined by the investigator according to RECIST v1.1 or death from any cause at 6 and 12 months. PD was defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum of diameters at prior timepoints (including baseline), in addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. K-M method was used to estimate PFS rate. Percentages have been rounded off. The event free rate used the K-M approach to estimate, which accounts for the censoring, the specific nature of time-to-event data. Naive calculation based on patient proportion will introduce bias.
Time Frame: Month 6, Month 12
Population: FAS included all randomized participants whether or not the participants received the assigned study treatment. Overall number analyzed is the number of participants with data available for analysis. Number analyzed is the number of participants with data available at the specified timepoint.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo + Atezolizumab + Carboplatin + Etoposide | Tiragolumab + Atezolizumab + Carboplatin + Etoposide
Number analyzed (Participants) | 23 | 28
percentage of participants
  Month 6 | 38.52 [26.20 to 50.84] | 46.71 [34.08 to 59.33]
  Month 12: number analyzed (Participants) | 7 | 15
  Month 12 | 12.70 [4.09 to 21.31] | 26.06 [14.84 to 37.29]
Statistical Analysis 1: Comparison: Placebo + Atezolizumab + Carboplatin + Etoposide vs Tiragolumab + Atezolizumab + Carboplatin + Etoposide; 6 Months; Test type: Superiority; p = 0.3633, Z-test; Difference in EFR at Month 6 = 8.18, 95% CI 2-sided [-9.46 to 25.82]
Statistical Analysis 2: Comparison: Placebo + Atezolizumab + Carboplatin + Etoposide vs Tiragolumab + Atezolizumab + Carboplatin + Etoposide; 12 Months; Test type: Superiority; p = 0.0642, Z-test; Difference in EFR at Month12 = 13.36, 95% CI 2-sided [-0.79 to 27.51]

11. Secondary Outcome: Overall Survival Rate at 12 Months and 24 Months in the PAS
Description: OS was defined as the time from the date of randomization to the date of death from any cause. OS rate at 12 months and 24 months was defined as the percentage of participants who did not experience death from any cause at 12 months and 24 months. Percentages have been rounded off.
Time Frame: Month 12, Month 24
Population: PAS included all randomized participants without presence or history of brain metastases at baseline. Overall number of participants analyzed is the number of participants with data available for analyses. Number analyzed is the number of participants with data available at the specified timepoint.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo + Atezolizumab + Carboplatin + Etoposide | Tiragolumab + Atezolizumab + Carboplatin + Etoposide
Number analyzed (Participants) | 27 | 38
percentage of participants
  Month 12 | 51.50 [38.09 to 64.92] | 71.97 [59.92 to 84.02]
  Month 24: number analyzed (Participants) | 13 | 15
  Month 24 | 32.94 [19.97 to 45.92] | 32.44 [19.55 to 45.33]
Statistical Analysis 1: Comparison: Placebo + Atezolizumab + Carboplatin + Etoposide vs Tiragolumab + Atezolizumab + Carboplatin + Etoposide; 12 Months; Test type: Superiority; p = 0.0261, Z-test; Difference in EFR = 20.47, 95% CI 2-sided [2.43 to 38.50]
Statistical Analysis 2: Comparison: Placebo + Atezolizumab + Carboplatin + Etoposide vs Tiragolumab + Atezolizumab + Carboplatin + Etoposide; 24 Months; Test type: Superiority; p = 0.9572, Z-test; Difference in EFR = -0.50, 95% CI 2-sided [-18.79 to 17.79]

12. Secondary Outcome: Overall Survival Rates at 12 Months and 24 Months in the FAS
Description: as for outcome 11
Time Frame: Month 12, Month 24
Population: FAS included all randomized participants whether or not the participants received the assigned study treatment. Overall number of participants analyzed is the number of participants with data available for analyses. Number analyzed is the number of participants with data available at the specified timepoint.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo + Atezolizumab + Carboplatin + Etoposide | Tiragolumab + Atezolizumab + Carboplatin + Etoposide
Number analyzed (Participants) | 32 | 41
percentage of participants
  12 Months | 54.73 [42.07 to 67.39] | 68.61 [56.91 to 80.32]
  24 Months: number analyzed (Participants) | 16 | 17
  24 Months | 34.65 [22.24 to 47.05] | 32.11 [20.06 to 44.16]
Statistical Analysis 1: Comparison: Placebo + Atezolizumab + Carboplatin + Etoposide vs Tiragolumab + Atezolizumab + Carboplatin + Etoposide; 12 Months; Test type: Superiority; p = 0.1145, Z-test; Difference in EFR = 13.88, 95% CI 2-sided [-3.36 to 31.12]
Statistical Analysis 2: Comparison: Placebo + Atezolizumab + Carboplatin + Etoposide vs Tiragolumab + Atezolizumab + Carboplatin + Etoposide; 24 Months; Test type: Superiority; p = 0.7734, Z-test; Difference in EFR = -2.54, 95% CI 2-sided [-19.83 to 14.75]

13. Secondary Outcome: Percentage of Participants With Adverse Events
Description: An AE is any untoward medical occurrence in a clinical investigation participant administered a pharmaceutical product, regardless of causal attribution. An adverse event can therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product, any new disease or exacerbation of an existing disease (a worsening in the character, frequency, or severity of a known condition), recurrence of an intermittent medical condition not present at baseline, any deterioration in a laboratory value or other clinical test that is associated with symptoms or leads to a change in study treatment or concomitant treatment or discontinuation from study drug or adverse events that are related to a protocol-mandated intervention, including those that occur prior to assignment of study treatment.
Time Frame: Up to 66 months
Reporting Status: Not Posted, anticipated posting 2026-04

14. Secondary Outcome: Time to Confirmed Deterioration (TTCD) Assessed Using European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire-Core (QLQ-C30) Score in the PAS
Time Frame: Up to approximately 66 months
Reporting Status: Not Posted, anticipated posting 2026-04

15. Secondary Outcome: TTCD Assessed Using EORTC QLQ-C30 Score in the FAS
Time Frame: Up to approximately 66 months
Reporting Status: Not Posted, anticipated posting 2026-04

16. Secondary Outcome: Maximum Plasma Concentration (Cmax) of Tiragolumab
Description: Only sparse pharmacokinetic samples were collected in this study. With the focus on only Cmax and Cmin, there are no additional PK timepoints not reported
Time Frame: Cycle 1 Day 1, 30 mins post end of infusion (EOI) (cycle length= 21 days)
Population: PK-evaluable population included all participants who received at least one dose of tiragolumab treatment and who have at least one post-baseline PK sample available.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram per milliliter (μg/mL)
Arm/Group | Tiragolumab + Atezolizumab + Carboplatin + Etoposide
Number analyzed (Participants) | 60
microgram per milliliter (μg/mL) | 175 (19.3)

17. Secondary Outcome: Minimum Plasma Concentration (Cmin) of Tiragolumab
Time Frame: Pre-dose, Day 1 of Cycles 2, 3, 4, 8, 12, 16 (cycle length= 21 days)
Population: PK-evaluable population included all participants who received at least one dose of tiragolumab treatment and who have at least one post-baseline PK sample available. Overall number of participants analyzed is the number of participants with data available for analyses. Number analyzed is the number of participants with data available for analyses at the specified timepoints.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | Tiragolumab + Atezolizumab + Carboplatin + Etoposide
Number analyzed (Participants) | 57
μg/mL
  Pre-dose: Cycle 2 Day 1 | 27.0 (51.6)
  Pre-dose: Cycle 3 Day 1: number analyzed (Participants) | 56
  Pre-dose: Cycle 3 Day 1 | 39.4 (79.9)
  Pre-dose: Cycle 4 Day 1: number analyzed (Participants) | 55
  Pre-dose: Cycle 4 Day 1 | 48.0 (40.0)
  Pre-dose: Cycle 8 Day 1: number analyzed (Participants) | 35
  Pre-dose: Cycle 8 Day 1 | 64.5 (44.7)
  Pre-dose: Cycle 12 Day 1: number analyzed (Participants) | 17
  Pre-dose: Cycle 12 Day 1 | 53.6 (193)
  Pre-dose: Cycle 16 Day 1: number analyzed (Participants) | 12
  Pre-dose: Cycle 16 Day 1 | 71.9 (58.8)

18. Secondary Outcome: Cmax of Atezolizumab
Time Frame: Cycle 1 Day 1, 30 mins post EOI (cycle length= 21 days)
Population: Atezolizumab PK evaluable set included all participants who received at least one dose of atezolizumab treatment and who have at least one post-baseline PK sample available.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram per milliliter (μg/mL)
Arm/Group | Placebo + Atezolizumab + Carboplatin + Etoposide | Tiragolumab + Atezolizumab + Carboplatin + Etoposide
Number analyzed (Participants) | 63 | 60
microgram per milliliter (μg/mL) | 355 (28.9) | 370 (36.5)

19. Secondary Outcome: Cmin of Atezolizumab
Time Frame: Pre-dose, Day 1 of Cycles 2, 3, 4, 8, 12, 16 (cycle length= 21 days)
Population: Atezolizumab PK evaluable set included all participants who received at least one dose of atezolizumab treatment and who have at least one post-baseline PK sample available. Overall number of participants analyzed is the number of participants with data available for analyses. Number analyzed is the number of participants with data available for analyses at the specified timepoints.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | Tiragolumab + Atezolizumab + Carboplatin + Etoposide | Placebo + Atezolizumab + Carboplatin + Etoposide
Number analyzed (Participants) | 57 | 58
μg/mL
  Pre-dose: Cycle 2 Day 1 | 63.8 (76.5) | 68.1 (33.7)
  Pre-dose: Cycle 3 Day 1: number analyzed (Participants) | 56 | 53
  Pre-dose: Cycle 3 Day 1 | 88.5 (166) | 96.6 (46.6)
  Pre-dose: Cycle 4 Day 1: number analyzed (Participants) | 55 | 53
  Pre-dose: Cycle 4 Day 1 | 111 (88.6) | 99.2 (62.7)
  Pre-dose: Cycle 8 Day 1: number analyzed (Participants) | 35 | 32
  Pre-dose: Cycle 8 Day 1 | 151 (41.6) | 151 (31.8)
  Pre-dose: Cycle 12 Day 1: number analyzed (Participants) | 17 | 14
  Pre-dose: Cycle 12 Day 1 | 139 (155) | 172 (35.0)
  Pre-dose: Cycle 16 Day 1: number analyzed (Participants) | 12 | 7
  Pre-dose: Cycle 16 Day 1 | 177 (55.0) | 169 (30.1)

20. Secondary Outcome: Percentage of Participants With Anti-Drug Antibodies (ADAs) to Tiragolumab
Time Frame: Predose on Day 1 of Cycles (each cycle=21 days) 1, 2, 3, 4, 8, 12, 16 and at TD visit (up to approximately 49 months)
Reporting Status: Not Posted, anticipated posting 2026-04

ADVERSE EVENTS:
Time Frame: Up to 32.3 months
Description: Safety population included all participants who received at least one dose of the study drug. One participant from the tiragolumab arm did not receive tiragolumab and hence was included in the placebo arm group for safety analysis. AEs collected up to the primary completion date are reported here. Adverse events section will be updated one year after the study completion date.
Arm/Group | Placebo + Atezolizumab + Carboplatin + Etoposide | Tiragolumab + Atezolizumab + Carboplatin + Etoposide
All-Cause Mortality (participants affected / at risk) | 40/63 | 43/60
Serious Adverse Events (participants affected / at risk) | 23/63 | 21/60
Other Adverse Events (participants affected / at risk) | 60/63 | 60/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo + Atezolizumab + Carboplatin + Etoposide (N=63) | Tiragolumab + Atezolizumab + Carboplatin + Etoposide (N=60)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Myelosuppression (Blood and lymphatic system disorders) | 4 (4) | 3 (3)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Cardiac failure (Cardiac disorders) | 2 (2) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 1 (1)
Goitre (Endocrine disorders) | 0 (0) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal polyp (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 2 (2)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 2 (2)
Infective exacerbation of bronchiectasis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 4 (4)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Skull fractured base (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 3 (3) | 1 (1)
Platelet count decreased (Investigations) | 3 (3) | 5 (5)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (2) | 2 (2)
Ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Immune-mediated lung disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory tract haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dermatitis exfoliative (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pelvic venous thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Vena cava thrombosis (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo + Atezolizumab + Carboplatin + Etoposide (N=63) | Tiragolumab + Atezolizumab + Carboplatin + Etoposide (N=60)
Anaemia (Blood and lymphatic system disorders) | 56 (100) | 58 (122)
Leukopenia (Blood and lymphatic system disorders) | 10 (25) | 10 (29)
Neutropenia (Blood and lymphatic system disorders) | 8 (21) | 13 (30)
Thrombocytopenia (Blood and lymphatic system disorders) | 6 (10) | 9 (15)
Atrial fibrillation (Cardiac disorders) | 4 (4) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 3 (4) | 4 (7)
Supraventricular extrasystoles (Cardiac disorders) | 0 (0) | 4 (4)
Hyperthyroidism (Endocrine disorders) | 3 (3) | 3 (4)
Hypothyroidism (Endocrine disorders) | 7 (7) | 6 (8)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 4 (4)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 3 (3)
Constipation (Gastrointestinal disorders) | 19 (24) | 17 (19)
Diarrhoea (Gastrointestinal disorders) | 5 (6) | 5 (6)
Nausea (Gastrointestinal disorders) | 13 (17) | 15 (23)
Toothache (Gastrointestinal disorders) | 1 (1) | 3 (3)
Vomiting (Gastrointestinal disorders) | 9 (9) | 10 (12)
Asthenia (General disorders) | 4 (5) | 4 (4)
Chest discomfort (General disorders) | 1 (1) | 3 (3)
Chest pain (General disorders) | 3 (3) | 3 (3)
Fatigue (General disorders) | 3 (3) | 10 (12)
Influenza like illness (General disorders) | 0 (0) | 3 (4)
Malaise (General disorders) | 4 (4) | 7 (7)
Oedema peripheral (General disorders) | 0 (0) | 3 (3)
Pain (General disorders) | 3 (3) | 3 (3)
Pyrexia (General disorders) | 10 (11) | 10 (13)
Pneumonia (Infections and infestations) | 9 (9) | 3 (3)
Infusion related reaction (Injury, poisoning and procedural complications) | 4 (4) | 10 (15)
Alanine aminotransferase increased (Investigations) | 18 (30) | 19 (37)
Aspartate aminotransferase increased (Investigations) | 18 (25) | 14 (31)
Bilirubin conjugated increased (Investigations) | 4 (7) | 4 (5)
Blood alkaline phosphatase increased (Investigations) | 7 (8) | 7 (11)
Blood bilirubin increased (Investigations) | 4 (12) | 5 (9)
Blood creatine phosphokinase increased (Investigations) | 4 (8) | 4 (4)
Blood creatinine increased (Investigations) | 2 (3) | 4 (5)
Blood lactate dehydrogenase increased (Investigations) | 9 (13) | 12 (16)
Blood thyroid stimulating hormone increased (Investigations) | 3 (3) | 4 (4)
Blood uric acid increased (Investigations) | 2 (3) | 3 (3)
Electrocardiogram QT prolonged (Investigations) | 3 (4) | 4 (9)
Gamma-glutamyltransferase increased (Investigations) | 10 (13) | 8 (13)
Lymphocyte count decreased (Investigations) | 6 (12) | 7 (37)
Neutrophil count decreased (Investigations) | 42 (101) | 44 (144)
Platelet count decreased (Investigations) | 40 (99) | 39 (134)
Weight decreased (Investigations) | 12 (13) | 9 (9)
Weight increased (Investigations) | 4 (5) | 6 (6)
White blood cell count decreased (Investigations) | 42 (105) | 42 (144)
Decreased appetite (Metabolism and nutrition disorders) | 14 (16) | 13 (15)
Hyperglycaemia (Metabolism and nutrition disorders) | 8 (13) | 6 (7)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 4 (5) | 4 (4)
Hyperuricaemia (Metabolism and nutrition disorders) | 8 (14) | 11 (15)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 16 (26) | 13 (31)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (2) | 4 (12)
Hypochloraemia (Metabolism and nutrition disorders) | 2 (2) | 4 (6)
Hypokalaemia (Metabolism and nutrition disorders) | 5 (7) | 7 (9)
Hypomagnesaemia (Metabolism and nutrition disorders) | 3 (4) | 4 (6)
Hyponatraemia (Metabolism and nutrition disorders) | 19 (27) | 15 (20)
Hypophosphataemia (Metabolism and nutrition disorders) | 4 (4) | 5 (10)
Hypoproteinaemia (Metabolism and nutrition disorders) | 1 (1) | 4 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 6 (6)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4)
Insomnia (Psychiatric disorders) | 4 (6) | 6 (7)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (8) | 12 (14)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 8 (8) | 21 (21)
Pruritus (Skin and subcutaneous tissue disorders) | 6 (6) | 10 (14)
Rash (Skin and subcutaneous tissue disorders) | 9 (10) | 17 (25)
Hypertension (Vascular disorders) | 1 (1) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2023-12-14): https://cdn.clinicaltrials.gov/large-docs/56/NCT04665856/Prot_000.pdf
  • Statistical Analysis Plan (2022-05-27): https://cdn.clinicaltrials.gov/large-docs/56/NCT04665856/SAP_001.pdf